CLINICAL TRIAL: NCT06915792
Title: Postpartum Evaluation of Antihypertensive Cessation and Efficacy (PEACE): A Randomized Controlled Trial Comparing Oral Labetalol and Oral Extended-Release Nifedipine for Managing Postpartum Hypertension
Brief Title: PEACE Trial: Postpartum Evaluation of Antihypertensive Cessation and Efficacy
Acronym: PEACE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tina A. Nguyen, MD, Associate Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-6051
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Hypertension (PPHT)
Keywords: postpartum hypertension, blood pressure control, labetalol, nifedipine, antihypertensive therapy, pregnancy hypertension, maternal health, randomized controlled
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Labetalol; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Labetalol (Experimental): Participants in this arm will receive oral labetalol to manage postpartum hypertension. The starting dose will be 200 mg twice or three times daily (BID or TID), with adjustments up to 2400 mg/day (800 mg TID) as needed.
  Interventions: Drug: Labetalol
- Nifedipine (Experimental): Participants in this arm will receive oral extended-release nifedipine to manage postpartum hypertension. The starting dose will be 30 mg once daily, with adjustments up to 120 mg/day as needed
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Labetalol — Labetalol is a beta-blocker commonly used to manage hypertension in pregnancy and postpartum. In this study, oral labetalol will be initiated at 200mg twice or three times daily and adjusted up to 2400 mg/day as needed for blood pressure control.
  Arms: Labetalol
Drug: Nifedipine — Nifedipine is a calcium channel blocker commonly used to manage hypertension in pregnancy and postpartum. In this study, oral extended-release nifedipine will be initiated at 30mg once daily and adjusted up to 120mg/day as needed for blood pressure control.
  Arms: Nifedipine

SUMMARY:
This randomized controlled trial compares two common medications, labetalol and extended-release nifedipine, to determine which is more effective at managing postpartum high blood pressure. We hypothesize that extended-release nifedipine will better control blood pressure and reduce the need for continued medication beyond six weeks postpartum. The study will enroll 110 postpartum participants, randomly assigning them to one of the two medications, with remote blood pressure monitoring to evaluate treatment effectiveness and inform postpartum hypertension management.

DETAILED DESCRIPTION:
Hypertensive disorders complicate approximately 10% of pregnancies in the United States and are among the leading causes of maternal morbidity and mortality worldwide. These conditions often emerge or persist after delivery, leading to postpartum hypertension. Postpartum hypertension has been associated with the development of chronic hypertension and other cardiovascular concerns, as well as risk of severe complications such as stroke and seizure, and represents a substantial reason for hospital readmission. While oral labetalol and oral extended-release nifedipine are the most commonly prescribed antihypertensive medications, there is limited evidence comparing their efficacy in managing postpartum hypertension. This study aims to address this gap by evaluating the outcomes of these medications on sustained blood pressure control in the postpartum period.

This prospective randomized controlled trial plans to enroll 110 participants with 55 individuals randomized to receive either oral labetalol or oral extended-release nifedipine. The primary outcome is continuation of antihypertensive medication beyond 6 weeks postpartum. Secondary outcomes include postpartum hospital readmission, medication side effects, and medication failure, defined as the need to switch the study medication or to add a second antihypertensive agent.

The study population will consist of postpartum adults with hypertensive disorders of pregnancy admitted at a tertiary care center, Ronald Reagan UCLA Medical Center, following delivery at ≥28 weeks gestation. Eligible individuals will have elevated postpartum blood pressures requiring initiation of an oral antihypertensive medication during their postpartum hospital stay or within 7 days of discharge. Individuals who have been treated with oral antihypertensive medication prior to delivery, contraindications to nifedipine or labetalol, or severe comorbidities will be excluded. On discharge, participants will be enrolled in remote blood pressure monitoring; blood pressure logs will be monitored daily by a dedicated nurse and overseen by a maternal-fetal medicine specialist who will make any necessary medication adjustments. Apart from random assignment of the study medication, all postpartum care will proceed as usual according to the study institution's standard clinical protocols.

This study is designed to provide evidence to inform clinical guidelines that address the clinical needs of high-risk patients, potentially reducing maternal morbidity and improving care. Participation is voluntary, with informed consent obtained prior to enrollment. Close monitoring through remote monitoring and follow-up visits with the research team and primary obstetrician will ensure participant safety throughout the study.

ELIGIBILITY:
Inclusion criteria:

Age ≥18 years Delivery at study institution at ≥28 weeks gestation Postpartum SBP > 150 and/or DBP > 100 OR 2 or more SBP > 140 and/or DBP > 90 within a 24-hour period Require initiation of an oral antihypertensive medication during postpartum hospital stay or within 7 days of discharge Treating obstetric team amenable to starting either study medication

Exclusion criteria:

Treated with oral antihypertensive medications prior to delivery Known allergies or contraindications to nifedipine or labetalol History of moderate persistent to severe asthma, chronic obstructive pulmonary disease, heart failure, or greater than first-degree atrioventricular heart block Unable to provide written informed consent in English

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Continuation of antihypertensive medication | 6 week postpartum
  The proportion of participants who continue to require antihypertensive medication beyond 6 weeks postpartum

SECONDARY OUTCOMES:
Postpartum hospital readmission | 6 weeks postpartum
  The number of participants requiring hospital readmission for hypertension-related complications.
Treatment failure | 6 weeks postpartum
  The proportion of participants requiring a medication switch or the addition of a second antihypertensive agent to achieve blood pressure control.
Patient-reported medication side effects | 6 weeks postpartum
  The frequency and type of medication-related side effects reported by participants.

IPD SHARING:
Plan to Share IPD: No